CLINICAL TRIAL: NCT06169176
Title: Intermediate-Size Expanded Access Trial of Autologous Hybrid TREG /Th2 T Stem Cell Therapy (RAPA-501) of Amyotrophic Lateral Sclerosis
Brief Title: RAPA-501 Therapy of ALS Expanded Access Protocol
Status: Temporarily not available | Type: Expanded Access
Sponsor: Rapa Therapeutics LLC (Industry)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: RAPA-501-ALS-EAP; 1U01NS136020-01 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; RAPA-501; ALS; Autologous TREG/Th2 T stem cell therapy; Rare Disease; Orphan Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Rare Diseases

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Other: RAPA-501 Autologous T stem cells — Experimental: Intermediate size expanded access cohort. Single-agent RAPA-501 T stem cells, (80 x 10EE6 cells per infusion; acceptable dose range of RAPA-501 T stem cells is 20-to-80 x 10EE6 cells per infusion.

SUMMARY:
RAPA-501-ALS is an Intermediate-Size Expanded Access Trial of RAPA-501 autologous hybrid TREG/Th2 T stem cells in patients living with amyotrophic lateral sclerosis (pwALS).

DETAILED DESCRIPTION:
ALS is a rare disease that is considered an orphan disease according to the Orphan Drug Act.

This is an open-label, non-randomized, multi-center intermediate size expanded access clinical trial of single-agent RAPA-501 T stem cells in patients with high-risk ALS who are not eligible for other ALS clinical trials.

After a subject consents to the study, an apheresis procedure will be performed to collect cells to manufacture the investigational product, RAPA-501 T stem cells. RAPA-501 cells are manufactured ex vivo using epigenetic reprogramming to yield a T stem cell population that is enriched for a dual anti-inflammatory phenotype based on hybrid TREG and Th2 differentiation. RAPA-501 T stem cells express both the TREG and Th2 transcription factors FOXP3 and GATA3, are enriched for expression of the ATP ectonucleotidase molecules CD39 and CD73, are enriched for the T cell homing molecule CD103, and suppress both effector T cell inflammatory molecules and CNS microglial cell inflammatory molecules.

This study is evaluating RAPA-501 T stem cell therapy at the dose of 80 x 10EE6 cells per infusion, with up to 4 infusions separated by six weeks between doses (infusion at time 0, and then after week 6, 12, and 18). Study subjects are then followed for several months to capture major clinical events and to assess survival. The total duration of RAPA-501 T stem cell therapy and follow-up interval on this protocol is approximately 8-months (250 days). The primary objective in the expanded access cohort is to determine the feasibility and safety of the highest-dose established safe dose of RAPA-501 (80 x 10EE6 cells per infusion). Secondary study objectives relate to assessment of overall survival compared to historical controls and determining the ALS disease activity pre-therapy, during study interventions, and throughout the post-therapy observation interval of RAPA-501 therapy through the monitoring of ALSFRS-R scores, SVC values, hand grip strength, and ROADS Scale. In addition, secondary study objectives relate to characterizing immune system parameters pre- and post- therapy and the potential effect of RAPA-501 therapy on serum markers of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Patients with sporadic or familial ALS diagnosed as laboratory-supported possible, probable, or definite according to World Federation of Neurology El Escorial Criteria.
3. Pulmonary slow vital capacity (SVC) < 50% of predicted normal (as measured within three months prior to screening or at the time of screening; inability to measure an SVC value at the time of screening that is due to severe reduction in respiratory function will also fulfill this eligibility criterion #3). However, SVC values ≥50% are acceptable if an EAP recipient of RAPA-501 is re-enrolled to the study.
4. Must have a source of autologous T cells potentially sufficient to manufacture RAPA-501 cells, as defined by a peripheral CD3+ T cell count ≥ 500 cells per μl.
5. Patients who are taking riluzole (Rilutek®), edaravone (Radicava®), and/or sodium phenylbutyrate/taurursodial (Relyvrio™) are eligible if taking the drug for at least 30 days prior to the screening visit.
6. Patients must be ≥ two (2) weeks removed from major surgery, or investigational therapy.
7. Patients must have no ongoing, unstable serious illness other than ALS, as determined by the Site Investigator.
8. Serum creatinine less than or equal to 2.0 mg/dL.
9. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN).
10. Bilirubin ≤ 1.5 (except if due to Gilbert's disease).
11. No history of abnormal bleeding tendency.
12. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future care.
13. Not enrolled in another interventional clinical trial or expanded access protocol and must have stopped taking other experimental drug(s) at least 2 weeks prior to screening.

Exclusion Criteria:

1. Active uncontrolled infection.
2. Hypertension not adequately controlled by ≤ 3 medications.
3. History of documented pulmonary embolus within 6 months of enrollment.
4. Clinically significant cardiac pathology, as defined by: myocardial infarction within 6 months prior to enrollment, Class III or IV heart failure according to NYHA, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
5. HIV, hepatitis B, or hepatitis C seropositive.
6. Pregnant or breastfeeding subjects.
7. Subjects of childbearing age, or males who have a partner of childbearing potential, who are unwilling to practice contraception.
8. Subjects may be excluded at the Principal Investigator discretion or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Fowler, M.D., Study Director — Rapa Therapeutics LLC
Locations (10):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Hospital Phoenix, Scottsdale, Arizona
  - University of California Irvine Health, Irvine, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Providence Portland Medical Center, Portland, Oregon